CLINICAL TRIAL: NCT04491227
Title: Global Assessment of Acute and Chronic Kidney Disease Incidence and Outcomes in Patients With COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ravindra Mehta, Recall Faculty, University of California, San Diego
Other Study IDs: 000295
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Covid19; AKI; CKD; ESRD; Transplant;Failure,Kidney
Keywords: AKI; dialysis; CKD; COVID19; renal transplant; mortality; renal recovery; resource utilization
MeSH Terms: conditions — COVID-19; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney disease in COVID-19: Chronic Kidney Disease (CKD): Known diagnosis of chronic kidney disease; prior evidence of markers of kidney damage for 3 months (microalbuminuria, proteinuria >300mg/24 hrs or abnormalities in imaging tests) or the presence of glomerular filtration rate (GFR) <60 mL/min/1.73 m2 for 3 months calculated with CKD-EPI equation, with or without other signs of kidney damage as described above.
  ESKD: Patients that are dialysis dependent.
  Suspected AKI: Oliguria (<200 mL/6 hours) and any AKI-related clinical signs or symptoms (see table 1) or urinalysis/dipstick abnormality. All suspected AKI cases must be confirmed prior to enrollment.
  Confirmed AKI: Meeting of at least one of the modified KDIGO Criteria
  * Increase or decrease in serum creatinine >0.3 mg/dl from reference in 48 hours
  * Increase or decrease in serum creatinine > 50% from reference in 7 days
  * Urine output < 400 ml/day
  Functioning Kidney transplant:

SUMMARY:
The coronavirus (COVID-19) pandemic has created a significant strain on health care resources across the world for managing critically ill patients. Emerging reports from China, South Korea and Italy have reported varying incidence of acute kidney (AKI) ranging from 5-15% with a mortality of 60-80% however there is no systematic assessment of the risk factors, recognition, course and outcomes in patients with and without kidney disease whose course is complicated by AKI1-4. Patients with underlying CKD, immunosuppressed patients with renal transplants and ESKD patients are at high risk for COVID-19 infection and there is limited information on the effect of COVID-19 on the course and outcomes of these patients. The requirement for renal support including IHD, CRRT and sorbent based therapies has been variable and has contributed to the intense pressure on the nephrology and critical care providers for delivering these therapies. As the COVID-19 pandemic expands in the USA and abroad, there is an intense need to understand the epidemiology of the disease and the resources needed for renal support to inform clinical management and public health interventions.

In this study, the investigators aim to investigate health care facilities across the world (hospital wards, ICU, outpatient clinics, nursing homes, healthcare centers) to draw a global picture of incidence, risk factors, resources available for treatment and prognosis of acute and chronic kidney disease in patient with COVID 19 confirmed infection. The aim is to identify trends in patients with acute and chronic kidney disease, determine its incidence, treatment and outcomes in different settings across the world. This information will be used to develop and implement educational tools and resources to prevent deaths from AKI and progression of CKD in this and following pandemics.

DETAILED DESCRIPTION:
Acute and Chronic kidney diseases are important causes of mortality and morbidity worldwide. The associated socioeconomic burden of kidney disease and AKI, as in some cases recovery is incomplete and chronic kidney disease (CKD) can arise, is a growing problem around the world. During the COVID 19 pandemic the incidence of AKI has been reported to be as low as 0.5% to as high as 23%. AKI was reported to develop at a median of 15 days in one study, and another study reported that most AKI developed within 7 days of admission. The data on acute kidney injury (AKI) in patients with COVID-19 is mostly from patients who are hospitalized, and in some studies limited to critically ill patients in the ICU. In ICU patients the requirement for renal support and mortality is reported to be high, however is a lack of epidemiological studies specifically designed to determine the impact of COVID 19 on kidney outcomes.

The mortality rate of patients with kidney dysfunction varies widely and is inversely related to country income and percentage of gross domestic product spent on total health expenditure. Several initiatives will be very insightful and identified important gaps in knowledge, more effort is required to understand this problem affecting all regions of the globe. In order to eventually implement resources and tools to help prevent, diagnose and treat patients with COVID 19 infection and kidney dysfunction, the investigators need to understand its incidence, risk factors, available resources and barriers to diagnosis and treatment.

This project will collect data on kidney function progression in patients infected with COVID 19 across the world. The study will open to individual physicians across the world who agreed to participate by providing de-identified clinical and lab data of patients with confirmed COVID 19 infection with acute and chronic kidney dysfunction.

Primary Objectives:

1. Establish incidence and outcomes of acute kidney injury (AKI) in different settings worldwide during the COVID 19 pandemic.

Secondary Objectives:

1. Compare risk factors, etiologies, diagnosis, management and outcomes of acute and chronic kidney dysfunction in COVID 19 patients in different countries
2. Determine resources available for recognition, non-dialytic and dialytic management and follow up of patients with acute and chronic kidney dysfunction and COVID 19 infection in different settings and countries.
3. Determine long term outcomes, 6 months and 1 year, of patients with acute and chronic kidney dysfunction and COVID 19 infection in different settings.
4. Evaluate barriers preventing access to the standard treatments of acute and chronic kidney dysfunction and COVID 19 infection across different countries.
5. Determine the impact of COVID 19 infection on the progression of acute and chronic kidney disease in patient with native and transplanted kidney.
6. Evaluate the treatment strategies of patient with ESKD on hospitalized patients with COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed infection with COVID 19
* Patients with Acute Kidney injury (AKI) or Chronic kidney disease (CKD) or need for dialysis
* Patients receiving Chronic dialysis (hemo or peritoneal dialysis)
* Renal transplant recipients

Exclusion Criteria:

* • Patients < 18 yrs age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID 19 infection with acute and chronic kidney dysfunction.
  Patients testing positive for COVID19 who meet criteria for AKI, have known CKD (with baseline eGFR less than 60), are ESKD on dialysis or kidney transplant recipients will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
AKI incidence | from hospital admission through hospital discharge upto 24 weeks
  Meeting of at least one of the modified KDIGO Criteria
  * Increase or decrease in serum creatinine >0.3 mg/dl from reference in 48 hours
  * Increase or decrease in serum creatinine > 50% from reference in 7 days
  * Urine output < 400 ml/day
Dialysis requirement | through study completion upto 1 year from enrollment
  initiation of intermittent hemodialysis, continuous hemodialysis or peritoneal dialysis during the hospital stay
hospital mortality | through study completion within 1 year
  Deaths during primary hospitalization

SECONDARY OUTCOMES:
Renal functional recovery | Assessed at at 3, 6 and 12 months from enrollment at hospital admission
  C-Complete: SCr < 0.3 mg/dL from reference P-Partial: Requires no dialysis but not complete recovery N-No recovery: Dialysis dependent C-Complete: SCr < 0.3 mg/dL from reference P-Partial: Requires no dialysis but not complete recovery N-No recovery: Dialysis dependent Percentage of patinets with renal functioanl recovery based on serum creatinien levels classfied as C-Complete: SCr < 0.3 mg/dL from reference P-Partial: Requires no dialysis but not complete recovery N-No recovery: Dialysis dependent
Functional status | questionnaires to be completed at 3, 6 and 12 months from enrollment at hospital admission
  EQL5D scale and SH8 scales completed at 3, 6 and 12 months post enrollment
Resource utilization | Within 1 year of enrollment for primary hospitalization
  Number of days patient is in the hospital and ICU and is managed with ventilators, dialysis or other extracorporeal organ support e.g. ECMO during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra L Mehta, Principal Investigator — University of California, San Diego
Locations (12):
- United States (5):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - University of Colorado, Aurora, Colorado
  - St. Peter's Hospital, Albany, New York
  - Jacobi Medical Center, New York, New York
- Hospital Obrero #2, Cochabamba, Bolivia
- Hopital Sacre Coeur & Universite de Montreal, Montreal, Quebec, Canada
- Universidad de Los Andes, Santiago, Chile
- Postgraduate Institute of Research, Chandigarh, Chandigarh, India
- United Kingdom (3):
  - Royal Free Hospital, London
  - Guy's & St Thomas's Hospital, London
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No
Participating sites will have acess to their own data and aggregate data